CLINICAL TRIAL: NCT02764281
Title: The Efficacy and Safety of Methotrexate, Etoposide, Dexamethasone and Pegaspargase Chemotherapy (MEDA) With Autologous HSCT in the Treatment of Stage IV Natural Killer/T-Cell Lymphoma: A Multicenter, Prospective Study
Brief Title: MEDA Chemotherapy and Autologous Hematopoietic Stem Cell Transplantation for Stage IV Natural Killer/T-cell Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Rong Tao, Dr, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1602
Record Dates: First submitted 2016-04-29; First posted 2016-05-06 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Extranodal NK-T-Cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Methotrexate; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEDA/Auto-HSCT (Experimental): Patients will be initially treated with four cycles MEDA chemotherapy, followed by autologous hematopoietic stem cell transplantation (Auto-HSCT).
  Interventions: Drug: MEDA; Procedure: Auto-HSCT

INTERVENTIONS:
Drug: MEDA — Methotrexate, 3.0g/m2/d iv, day 1
  Etoposide, 100mg/m2 iv, day 2 to day 4
  Dexamethasone, 40mg/d iv, day 1 to day 4
  Pegaspargase, 2500IU/m2/d im, day 4
  The MEDA chemotherapy will be repeated every 3 weeks.
  Other Names: Methotrexate, Etoposide,Dexamethasone,Pegaspargase
Procedure: Auto-HSCT — Auto-HSCT will be performed with patients who responded to the initial MEDA chemotherapy with standard BEAM conditioning regimen.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of methotrexate, etoposide, pegaspargase and dexamethasone (MEDA) chemotherapy and autologous hematopoietic stem cell transplantation (Auto-HSCT) in patients with stage IV extranodal natural killer/T-cell lymphoma, nasal type.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTCL), nasal type, is a rare subtype of non-Hodgkin lymphoma (NHL) with relatively high incidence in China. L-asparaginase based chemotherapy improved overall response and prolonged the long-term survival for patients with stage IV. But the optimal treatment schedule has not been established. This study is designed with four cycles MEDA chemotherapy, followed by Auto-HSCT for stage IV patients with newly onset, relapsed or refractory diseases. The efficacy and safety of this protocol in the treatment of will be measured.

ELIGIBILITY:
Inclusion Criteria:

Pathological diagnosis of extranodal natural killer/T-cell lymphoma, nasal type based on WHO 2008 classification of tumors of haematopoietic and lymphoid tissue.

Eastern Cooperative Oncology Group (ECOG ) performance status 0~3.

Stage IV disease with at least one measurable lesion.

Preserved organ functions for: Platelet>50×10*9/L, hemoglobin>80g/L, total bilirubin (TBIL)<3×ULN, alanine transaminase (ALT)<5×ULN, serum creatinine (Cr)<1.5×ULN, fibrinogen≥0.5g/L, LVEF≥50%.

Signed Informed consented.

Exclusion Criteria:

Relapsed or progressive disease to prior L-asparaginase-based chemotherapy.

Concurrent cancers need surgery or chemotherapy within 6 months.

History of chemotherapy or radiotherapy for other solid cancers within 3 years.

Recent history of radiotherapy of upper-aero-digestive tract within last 3 months.

Significant complications: LVEF≤50%, coagulopathy, autoimmune disease, severe infection, or liver cirrhosis, severe hemophagocytic lymphohistiocytosis.

Mental disorders.

Pregnant or lactation.

HIV, hepatitis virus C (HCV), or active hepatitis virus B (HBV) infection with HBV DNA≥10*5 copies/ml.

History of pancreatitis.

Known history for grade 3/4 allergy to the drugs in chemotherapy regimen.

Enrolled in other trial treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Complete response rate | Day 28 of the 4th course of MEDA chemotherapy
  The complete response rate will be assessed on day 28 of the 4th course of MEDA chemotherapy.

SECONDARY OUTCOMES:
Progression free survival | 2-year
  Progression free survival is the time from entry onto the treatment until lymphoma progression or death of any reason.
Overall response rate | Day 28 of the 4th course of MEDA chemotherapy
  The overall response rate will be assessed on day 28 of the 4th course of MEDA chemotherapy.
Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | Day 1 of each course of chemotherapy and then every 3 months for 2 years
  Treatment-Related Adverse Events will be assessed and graded by NCI CTCAE v4.0.
Overall survival | 2-year
  Overall survival is defiend as the time from entry onto the treatment until death of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Study Chair — Xinhua hospital, Shanghai Jiao Tong University of Medicine
Locations (7):
- China (7):
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Eye Ear Nose and Throat Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality
  - Shanghai Dong Fang hospital, Shanghai, Shanghai Municipality
  - Shanghai Tong Ren Hospital, Shanghai, Shanghai Municipality
  - Xin Jiang People's Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No